CLINICAL TRIAL: NCT06089798
Title: Analgesic Efficacy of Ultrasound-guided Bilateral Pecto-intercostal Fascial Block in Pediatric Cardiac Surgery
Brief Title: Analgesic Efficacy of Ultrasound-guided Bilateral Pecto-intercostal Plane Block in Pediatric Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Selin Saglam, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Other Study IDs: KAEK/2022.01.21
Record Dates: First submitted 2023-06-11; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Regional Anesthesia
Keywords: pecto-intercostal fascial block; pediatric congenital cardiac surgery; postoperative pain management

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PIFB Group: The patients in this group will be applied pecto-intercostal fascial block before surgical incision additional to general anesthesia.
- Nonblock Group: The patients in this group will be given only standard general anesthesia.

SUMMARY:
The goal of this study is to compare patients outcome in two groups. the first group will be applied pecto-intercostal fascial block additional to general anesthesia and the second group will not.

This is a single-center, prospective, observational trial to study the efficacy of Pecto-intercostal Fascial Block (PIFB) in patients undergoing pediatric congenital cardiac surgery requiring median sternotomy and cardiopulmonary bypass. The children are aged between 6 months to 12 years with American Society of Anesthesiologists (ASA) score 2 or 3.

The main question it aims to answer are:

The investigators' first question is if applying pecto-intercostal fascial block just after anesthesia induction reduces postoperative pain status. Secondly, if this pain status makes any reduction in preoperative opioid consumption. The investigators aim to find out; if there is any difference in opioid consumption during operation and postoperative 24-hour, postoperative Face, Legs, Activity, Cry, Consolability (FLACC) scale, length of intensive care unit and hospital stays, and other complications.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing pediatric congenital cardiac surgery requiring median sternotomy and cardiopulmonary bypass.
* age between 6 months and 12 years
* ASA score 2 or 3
* Risk Adjustment for Congenital Heart Surgery (RACHS-1) score under 4

Exclusion Criteria:

* patients who need mechanical ventilation support before surgery
* patients who need to stay intubated more than 24 hours after surgery
* patients undergo complex cardiac surgery with RACHS-1 score higher than 4.
* patients without consent
* having allergic reaction to bupivacaine
* having cardiac surgery before (redo patient)

Ages: 6 Months to 12 Years | Sex: All
Age Groups: Child
Study Population: Patients 6 months to 12 years old, undergoing pediatric congenital cardiac surgery requiring median sternotomy and cardiopulmonary bypass with ASA score 2 or 3.
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain Score | at the time of extubation, 1st hour after extubation, 2nd hour after extubation, 6th hour after extubation, 12th hour after extubation, 24th hour after extubation
  Face, Legs, Activity, Cry, Consolability scale (FLACC scale), FLACC is a behavioral pain assessment scale used for nonverbal or preverbal patients who are unable to self-report their level of pain. Pain is assessed through observation of 5 categories including face, legs, activity, cry, and consolability. The values are between 0 and 10. The higher the score the worse the pain and outcome.

SECONDARY OUTCOMES:
peroperative opioid consumption | during operation
  sum of fentanyl and remifentanil consumption in micrograms
Postoperative opioid consumption | From extubation to 24 hours after extubation.
  morphine usage in milligrams
dexmedetomidine consumption | From the beginning of dexmedetomidine infusion to 24 hours after extubation
  dexmedetomidine in micrograms
Paracetamol consumption | From extubation to 24 hours after extubation.
  paracetamol in milligrams

OTHER OUTCOMES:
extubation time | up to 24 hours
  time of extubation in hours
intensive care stay | up to 24 weeks
  length of intensive care stay in days
hospital stay | up to 1 year
  hospital stay in days

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Basaksehir, Turkey (Türkiye)